CLINICAL TRIAL: NCT02076945
Title: Characteristics of Popliteal Sciatic Nerve Block in Patients With and Without Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, MD; program director, regional aneshesia, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-40/14
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Neuropathy
Keywords: Regional anesthesia; Diabetic neuropathy; Ultrasound
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy patients (Active Comparator): Patients without diabetes and without peripheral neuropathy (based on the cross sectional area of the posterior tibial nerve 3 cm above the medial malleolus <19.01 mm2)
  Interventions: Procedure: US-guided sciatic block at the popliteal crease (30 mL1:1 mixture of lidocaine 1% and bupivacaine 0.5%)
- Diabetic patients without neuropathy (Experimental): Patients with diabetes but without peripheral neuropathy (based on the cross sectional area of the posterior tibial nerve 3 cm above the medial malleolus <19.01 mm2)
  Interventions: Procedure: US-guided sciatic block at the popliteal crease (30 mL1:1 mixture of lidocaine 1% and bupivacaine 0.5%)
- Diabetic patients with neuropathy (Experimental): Patients with diabetes and with peripheral neuropathy (based on the cross sectional area of the posterior tibial nerve 3 cm above the medial malleolus > 19.01 mm2)
  Interventions: Procedure: US-guided sciatic block at the popliteal crease (30 mL1:1 mixture of lidocaine 1% and bupivacaine 0.5%)

INTERVENTIONS:
Procedure: US-guided sciatic block at the popliteal crease (30 mL1:1 mixture of lidocaine 1% and bupivacaine 0.5%)

SUMMARY:
Background Between 25 and 55% of diabetic patients develop neuropathy secondary to hyperglycemia. High resolution bedside ultrasound has been demonstrated to be a useful tool to detect the presence of neuropathy prior to block performance, by measuring the cross-sectional area of the posterior tibial nerve: a value superior to 19.01 mm2 at a distance of 3 cm above the medial malleolus has an optimal threshold value for identification of diabetic sensorimotor polyneuropathy.

Animal data showed that duration of sciatic nerve block with local anesthetics is longer in diabetic rats compared with non-diabetic rats. Characteristics of a peripheral nerve blockade in humans with diabetic sensorimotor neuropathy are unknown.

Aim The aim of this study is to compare duration of analgesia and other characteristics of an ultrasound-guided popliteal sciatic nerve block between diabetic patients with neuropathy, diabetic patients without neuropathy and non-diabetic patients without neuropathy, based on the ultrasound-measured cross-sectional area of the posterior tibial nerve.

Hypothesis We hypothesize that diabetic patients with neuropathy will have a duration of analgesia lasting 50% longer than patients without neuropathy.

Methods This will be an observational study on diabetic and non-diabetic patients, with and without peripheral neuropathy, based on the ultrasound-measured cross sectional area of the posterior tibial nerve 3 cm above the medial malleolus (cut-off value, 19.01 mm2)

All patients will receive ultrasound-guided sciatic nerve block with 30 mL1:1 mixture of lidocaine 1% and bupivacaine 0.5%, with the needle tip positioned at the bifurcation of the sciatic nerve in peroneal and tibial nerve, below the common fascia or paraneurium. Block success will be confirmed by loss of sensation to pinprick in the distribution of the common peroneal and tibial nerves 30 minutes following local anesthetic injection. This procedure will be completed by a saphenous nerve block. Postoperative pain management will be standardized.

Pain and block-related endpoints will be collected such as onset time of action of sensory and motor blockades, duration of analgesia, pain scores and opiates consumption among others.

Relevance Defining the duration of analgesia in case of diabetic neuropathy will help regional anesthesiologists to better define the type and doses of drugs that will be injected and to better prescribe the postoperative multimodal analgesic treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-85 years old
* patients scheduled to undergo foot surgery

Exclusion Criteria

* patients with neuropathy caused by genetic, metabolic and inflammatory diseases, as well as toxic agents and drugs (eg chemotherapy agents);
* patients with chronic pain syndrome;
* patients with contraindications for regional anesthesia (e.g., allergy to local anesthetics);
* chronic consumption of opioids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | with 24 hours after block performance

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV (Centre Hospitalier Universitaire Vaudois), Lausanne, Canton of Vaud, Switzerland